CLINICAL TRIAL: NCT02312492
Title: Development of a Novel Method to Study in Vivo Fatty Acid Metabolism Using Stable Isotope Labeled Fatty Acids in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1542 - Fatty Acid Kinetics
Record Dates: First submitted 2014-06-04; First posted 2014-12-09 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dyslipidemia
Keywords: fatty acid kinetics
MeSH Terms: conditions — Dyslipidemias | interventions — Oleic Acid; Palmitic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 18:1 diet (Experimental): Oleic Diet - volunteers will consume oleic enriched food for a period of 5 weeks.
  Interventions: Other: Oleic Diet
- 16:0 diet (Experimental): Palmitic diet - Volunteers will consume palmitic enriched food for a period of 5 weeks.
  Interventions: Other: Palmitic Diet
- 18:0 (Experimental): Stearic Diet - Volunteers will receive Stearic enriched food for a period of 5 weeks.
  Interventions: Other: Stearic Diet

INTERVENTIONS:
Other: Oleic Diet — The 18:1 (oleic) diet will contain 55%E carbohydrate, 15%E protein, 30%E fat, 100 mg cholesterol/1000 kcal and 15 g fiber/1000 kcal. The vegetable oils and/or fats (henceforth collectively referred to as experimental oils) that will be used to formulate the diets were selected not only take into account the fatty acid of interest but also the fatty acid displaced within the context of an unchanged total fat content. This was accomplished by formulating a diet containing 10%E fat and then adding the experimental oils (oleic) to 30%E total fat by incorporating them into various food items intended for consumption throughout the day. The actual food items comprising the 3 diets will be similar, only differing in the experimental oils.
  Other Names: Diet enriched in oleic acid; 18:1
  Arms: 18:1 diet
Other: Palmitic Diet — The 16:0 (palmitic) diet will contain 55%E carbohydrate, 15%E protein, 30%E fat, 100 mg cholesterol/1000 kcal and 15 g fiber/1000 kcal. The vegetable oils and/or fats (henceforth collectively referred to as experimental oils) that will be used to formulate the diets were selected not only take into account the fatty acid of interest but also the fatty acid displaced within the context of an unchanged total fat content. This was accomplished by formulating a diet containing 10%E fat and then adding the experimental oils (palmitic) to 30%E total fat by incorporating them into various food items intended for consumption throughout the day. The actual food items comprising the 3 diets will be similar, only differing in the experimental oils.
  Other Names: Diet enriched in palmitic acid.; 16:0
  Arms: 16:0 diet
Other: Stearic Diet — The 18:0 diet (stearic) will contain 55%E carbohydrate, 15%E protein, 30%E fat, 100 mg cholesterol/1000 kcal and 15 g fiber/1000 kcal. The vegetable oils and/or fats (henceforth collectively referred to as experimental oils) that will be used to formulate the diets were selected not only take into account the fatty acid of interest but also the fatty acid displaced within the context of an unchanged total fat content. This was accomplished by formulating a diet containing 10%E fat and then adding the experimental oil (stearic) to 30%E total fat by incorporating them into various food items intended for consumption throughout the day. The actual food items comprising the 3 diets will be similar, only differing in the experimental oils.
  Other Names: Stearic acid enriched diet.; 18:0
  Arms: 18:0

SUMMARY:
Specific Aim 1: To compare the metabolic fate (transport, conversion and oxidation) of labeled 18:0 (13C18:0) and its metabolic product 18:1 (13C18:1) in the fed state after habituation to diets enriched in the corresponding fatty acid.

Hypothesis: In the fed state, the metabolic fate of 13C18:0 compared to 13C18:1 will be characterized by similar transport, higher conversion, and similar oxidation rates..

DETAILED DESCRIPTION:
Vegetable oils high in the specific fatty acids of interest - stearic (found in cocoa butter, meats), palmitic (found in meats, dairy and some plant oils) and stearic acid's metabolic product, oleic (found in olive and corn oil) - will be used to displace each other in a standardized diet and fed to mildly hypercholesterolemic postmenopausal women using a randomized-controlled crossover design. Six women who are enrolled in 10150 - Study A will be invited to participate in this study. Each of the phases will be 5 weeks in length with a 2-4 week break between phases. All food and drink will be provided to study volunteers. Blood pressure and body weight will be monitored once per week and adjustments made, if necessary, to maintain a stable weight. During week 1 of the 18:0 and 18:1 dietary phases, a fasting blood sample will be drawn. A single stool sample will be collected on any of the study visits after week three. On Day 1 of week 5, following a 12 hour fast, each volunteer will receive their usual diet divided into 15 hourly small meals. A purified tracer dose (1 mg/kg bodyweight [BW]) of 13C fatty acid will be incorporated into the 1pm meal. Blood samples will be collected from a catheter inserted into the subcubital vein just before consuming the first hourly meal and then 2, 5, 7, 8, 9, 11, 13 and 15 hours thereafter. Breath samples will be collected before the first hourly meal as well as at various time-points after. Additional fasting blood samples will be collected on Days 2, 3, 4 and 5 of the 18:0 and 18:1 diet phases. At the end of Day 1, volunteers will have the option of returning home or staying overnight at the Jean Mayer Human Nutrition Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (menopause defined by complete natural cessation of menses for >12 months or a bilateral oophorectomy).
* Age >50 to < 85 years
* BMI >20 to <35 kg/m2
* LDL-cholesterol >100 mg/dL
* CRP (C reactive protein) <10 ug/dL
* Normal fasting plasma glucose levels (<120 mg/dL)
* Not taking medication known to affect lipid metabolism:

HMG-CoA reductase inhibitors (statins)

* Bile Acid Sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.)
* Cholesterol Absorption Inhibitors (Ezetimibe [Zetia])
* Nicotinic Acid Agents (Niacin, Niacor, Slo-Niacin, etc)
* Fibrates (Gemfibrozil, Clofibrate, Ciprofibrate, Fenofibrate [Tricor], etc)
* Probucol
* Anticoagulants (Coumadin, Heparin, Plavix, etc)
* Hormone therapy medications containing estrogen
* Acetylsalicylic acid containing medications, aspirin
* Diphenylhydantoin
* Supplements containing fatty acids (Fish Oil, Flaxseed, etc.) and any other compounds that affect lipid metabolism (red yeast rice, etc.) for at least 3 months prior to participation in the study
* Anabolic steroids
* Hydrocortisone

  * Normal kidney function as assessed by serum creatinine and blood urea nitrogen
  * Normal liver function as assessed by serum glutamic pyruvic transaminase, serum glutamic oxaloacetic transaminase and alkaline phosphatase
  * Normal thyroid function as assessed by serum TSH (thyroid stimulating hormone)
  * Normal gastrointestinal function
  * Normotensive on or off medication
  * Non-smoker for at least 2 years
  * Alcohol intake < 7 drinks per week, and willingness to abstain from consuming alcohol while participating in the study.
  * Consistent physical activity
  * Willingness to follow protocol as detailed in the Institutional Review Board (IRB) approved consent form.

Exclusion Criteria:

* Men
* Women who have had a double mastectomy
* Age < 50 and > 85 years
* BMI < 20 and > 35 kg/m2
* LDL-cholesterol <100 mg/dL
* CRP > 10 ug/dL
* Abnormal fasting plasma glucose levels >120 mg/dL
* Use of medications known to affect lipid metabolism:

  * HMG-CoA reductase inhibitors (statins)
  * Bile Acid Sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.)
  * Cholesterol Absorption Inhibitors (Ezetimibe [Zetia])
  * Nicotinic Acid Agents (Niacin, Niacor, Slo-Niacin, etc)
  * Fibrates (Gemfibrozil, Clofibrate, Ciprofibrate, Fenofibrate [Tricor], etc)
  * Anticoagulants (Coumadin, Heparin, Plavix, etc)
  * Hormone therapy medications containing estrogen
  * Probucol
  * Acetylsalicylic acid containing medications, aspirin
  * Diphenylhydantoin
  * Supplements containing fatty acids (Fish Oil, Flaxseed, etc.) and any other compounds that affect lipid metabolism (red yeast rice, etc.) in the last 3 months prior to participation in the study
  * Anabolic steroids and hydrocortisone
* Renal or kidney disease, as defined by a history of chronic kidney disease or by glomerular filtration rate of < 60 ml.min/1.73 m2 calculated from screening blood tests.
* Hypothyroidism or hyperthyroidism, as defined as screening TSH outside of normal ranges (<0.4 or >4.5), unless controlled with medication for at least 6 months
* Gastrointestinal disease
* Uncontrolled hypertension or high BP reading at the discretion of the study physician or nurse
* Established cardiovascular disease as defined by history of myocardial infarction, stroke, heart failure, coronary artery bypass graft, stenosis >50%, angina and peripheral arterial disease)
* Anemia, as defined by screening haemoglobin <11.7g/dL.
* Liver disease, as defined by a history of chronic hepatitis B or C, cholestatic or cirrhotic liver disease, nonalcoholic fatty liver disease, elevations of SGPT or SGOT greater than 1.5 times the upper limit of normal at screening, bilirubin greater than 2 mg/dL (in the absence of benign causes of elevated bilirubin such as Gilbert's syndrome) at screening, or albumin below the lower limit of normal.
* Type I and II diabetes
* Any non-steroidal anti-inflammatory drugs (NSAID) or antihistamine use by subject for 72 hours prior to blood draws
* Smoking or use of nicotine-containing products within the past 2 years
* Alcohol intake > 7 drinks per week or unwillingness to abstain from consuming alcohol while participating in the study
* Unwillingness to maintain body weight during participation in the study
* Unwillingness to adhere to diet and study protocol
* Weight gain or loss of more than 15 lb within 6 months prior to enrollment
* Vegetarians and those with food allergies or aversions
* Non-English speaking subjects
* No Social Security number
* Women who have a history of difficulty with blood draws
* Blood donation within the past 8 weeks

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
fatty acid kinetics in total plasma | 15 weeks
  measurement of isotope ratio (13C:12C) in total plasma, cholesterol ester, triglyceride, phospholipid, monoglyceride and diglyceride subfractions as well as chylomicrons, VLDL (very low density lipoprotein), TRL (triglyceride-rich lipoprotein), LDL (low density lipoprotein) and HDL (high density lipoprotein).
fatty acid kinetics in cholesterol ester | 15 weeks
fatty acid kinetics in triglyceride | 15 weeks
fatty acid kinetics in phospholipid | 15 weeks
fatty acid kinetics in monoglyceride subfraction | 15 weeks
fatty acid kinetics in diglyceride subfraction | 15 weeks
fatty acid kinetics in chylomicrons | 15 weeks
fatty acid kinetics in VLDL (very low density lipoprotein) | 15 weeks
fatty acid kinetics in TRL (triglyceride-rich lipoprotein) | 15 weeks
fatty acid kinetics in LDL (low density lipoprotein) | 15 weeks
fatty acid kinetics in HDL (high density lipoprotein) | 15 weeks

SECONDARY OUTCOMES:
rate of oxidation | 15 weeks
  breath analysis will be conducted to determine rate of oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts University/HNRCA
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States